CLINICAL TRIAL: NCT01651325
Title: A Phase 1, Open-Label, Sequential Study of the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Dextromethorphan in Healthy Adult Subjects
Brief Title: Drug Interaction Study of Multiple Doses of Isavuconazole and Single Dose of Dextromethorphan in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0042
Record Dates: First submitted 2012-07-23; First posted 2012-07-27 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Dextromethorphan; Healthy Adult Volunteers
Keywords: Isavuconazole; dextromethorphan; dextrorphan; DXM; Healthy Volunteers; BAL4815
MeSH Terms: interventions — isavuconazole; Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and dextromethorphan (Experimental): Dextromethorphan on Day 1and Day 10, Isavuconazole three times per day (TID) on Days 6 and 7, and once daily (QD) on Days 8 thru 12.
  Interventions: Drug: Isavuconazole; Drug: dextromethorphan

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL4815; ASP9766
Drug: dextromethorphan — oral
  Other Names: DXM

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics of a single dose of dextromethorphan in healthy adult subjects.

DETAILED DESCRIPTION:
Subjects will check-in on Day -1 and remain confined to the clinical unit until Day 13. On the morning of Day 1, subjects will receive a single dose of dextromethorphan. On Days 6 and 7, subjects will receive isavuconazole three times daily (TID) administered approximately 8 hours apart. On Day 8 through 12, subjects will receive isavuconazole once daily (QD). On Day 10, subjects will receive a single dose of dextromethorphan. A follow-up visit will be scheduled on Day 21 (± 2 days).

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45.0 kg and has a body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive
* The subject's 12-lead electrocardiogram (ECG) is normal at Screening and Day -1 or, if abnormal, the abnormality is not clinically significant as determined by the investigator, including a QTcF of 430 msec or less for male or 450 msec or less for female subjects
* The subject's clinical laboratory test results at Screening and Day -1 are within normal limits unless the investigator considers the abnormality to be not clinically significant. Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be ≤ upper limit of normal, and total bilirubin must be ≤ 1.5 mg/dL
* The female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years at Screening without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests at Screening and Day -1
* The male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study

Exclusion Criteria:

* The subject has any clinically significant (as judged by the Investigator) disease history of the following systems: pulmonary, gastrointestinal, cardiovascular (including a history of clinically significant arrhythmia or clinically significant conduction delays on ECG), hepatic, neurological, psychiatric, renal, genitourinary, endocrine, metabolic, dermatologic, immunologic, hematologic, or malignancy excluding non melanoma skin cancer
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check in on Day -1
* The subject has received a vaccination within the last 30 days prior to study drug administration or plans to receive any vaccinations during the study or within 2 weeks after the last dose of study drug
* The subject has a positive result for hepatitis C antibodies or hepatitis B surface antigen at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products including dextromethorphan or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods (as judged by the investigator), or a history of severe anaphylactic reactions
* The subject has smoked (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of occasional use of acetaminophen up to 2 g/day
* The subject has received an experimental agent within 30 days or 5 half-lives, whichever is longer, prior to Day -1
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or has donated plasma within 7 days prior to clinic check-in on Day -1
* The subject has taken part in strenuous exercise within 3 days prior to study drug administration
* The subject anticipates an inability to abstain from caffeine or alcohol use for 48 hours prior to clinical check-in on Day -1 and throughout the duration of the study; or from grapefruit, Seville oranges, star fruit, or any products containing these items from 72 hours prior to clinic check-in on Day -1 and throughout the duration of the study
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, as defined by the investigator, or a positive drug and/or alcohol screen at Screening or Day -1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile for dextromethorphan (in plasma): AUCinf, Cmax , AUClast | Pre-dose on Days 1 and 10, and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48 and 72 hours post-dose
  Area under the concentration-time curve (AUC) from time 0 extrapolated to infinity (AUCinf), maximum concentration (Cmax), and AUC from time of dosing to the last quantifiable concentration (AUClast).

SECONDARY OUTCOMES:
PK profile for dextromethorphan (in plasma): t1/2, tmax, CL/F, and Vz/F | Pre-dose on Days 1 and 10, and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48 and 72 hours post-dose
  Apparent terminal elimination half-life (t1/2), time to attain Cmax (tmax), apparent body clearance after oral dosing (CL/F), and apparent volume of distribution (Vz/F)
PK profile for dextrorphan (in plasma): AUClast, AUCinf, Cmax, tmax, t1/2 | Pre-dose on Days 1 and 10, and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48 and 72 hours post-dose
PK Isavuconazole (in plasma): trough concentration (Ctrough) | Pre-dose on Days 8 and 12 and at 24 (Day 13) hours post-dose
PK profile for Isavuconazole (in plasma): AUCtau, Cmax, and tmax | Day 9 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12,16, 20 hours post-dose and Day 10 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, and 24 (Day 11) hours post-dose
  AUC during time interval between consecutive dosing (AUCtau)
Safety assessed by recording of adverse events, clinical laboratory evaluation, electrocardiograms (ECGs) and vital signs | Day 1 through Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel, Baltimore, Maryland, United States